CLINICAL TRIAL: NCT07001137
Title: Medication Reconciliation Process in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0014_CASA
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Medication Reconciliation; Patient Safety; Geriatrics; Hospital Readmission; Pharmaceutical Services; Transitions of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Patients who did not receive any medication reconciliation (CTM)
- Patients who received CTM only at hospital admission
- Patients who received CTM at both admission and discharge

SUMMARY:
This study looks at how reviewing and confirming a patient's medications during a hospital stay can help reduce problems after they go home. It focuses on patients aged 75 and older who were admitted to a short-stay geriatric unit. The researchers compared three groups:

* Patients who did not receive any medication reconciliation (CTM),
* Patients who received CTM only at hospital admission,
* Patients who received CTM at both admission and discharge.

The goal was to see if this process could lower the number of hospital readmissions, emergency room visits, and deaths within six months after discharge. The study is based on real data from a hospital in 2019 and was conducted by pharmacists and doctors working together.

ELIGIBILITY:
Inclusion Criteria:

- All patients admitted to the short-stay geriatric unit of Casanova Hospital Between January 1st and August 31st, 2019

Exclusion Criteria:

- Patients who were discharged and then readmitted to the short-stay unit after a brief transfer to another unit (e.g., surgery, internal medicine, or intensive care).

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: The study population consists of elderly patients aged 75 years and older who were hospitalized in the short-stay geriatric unit of Casanova Hospital between January 1 and August 31, 2019. These patients typically present with multiple chronic conditions and are often prescribed numerous medications (polymedicated), making them particularly vulnerable to medication errors during care transitions.
  The population is selected from a hospital-based, real-world clinical setting, and reflects a high-risk group for hospital readmission, emergency visits, and medication-related complications.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Number of hospital readmissions within six months following discharge from the short-stay geriatric unit | Six months after discharge from the short-stay geriatric unit

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France